CLINICAL TRIAL: NCT06087237
Title: The Efficacy of Pentoxifylline in Reducing Post-surgical Complications in Patients Undergoing Breast Cancer Surgery
Brief Title: The Efficacy of Using Pentoxifylline in Patients Undergoing Breast Cancer Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Omar Hamdy, Doctor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-147
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Post-Surgical Complication; Breast Cancer Surgery
Keywords: pain; wound healing; post-surgery; breast cancer
MeSH Terms: conditions — Pain; Breast Neoplasms | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pentoxifylline group (Experimental): Two 400 mg extended-release pentoxifylline oral tablets are administered 2 hours before surgery, then one tablet three times per day after surgery, and continue for four weeks after the surgery. Standard of care for pain management, including paracetamol 1g IV every 8 hours and Ketorolac 30 mg IV every 12 hours.
  Interventions: Drug: Pentoxifylline
- Control group (Active Comparator): Patients recieved the standard of care without pentoxifylline.
  Interventions: Drug: paracetamol +ketorolac

INTERVENTIONS:
Drug: Pentoxifylline — Two 400 mg extended-release pentoxifylline oral tablets are administered 2 hours before surgery, then one tablet three times per day after surgery, and continued for four weeks after the surgery.
  Standard of care for pain management, including paracetamol 1g IV every 8 hours and Ketorolac 30 mg IV every 12 hours.
  Other Names: Trental tablets 400mg
  Arms: Pentoxifylline group
Drug: paracetamol +ketorolac — Patients receive the usual treatment only:
  paracetamol 1g IV every 8 hours and Ketorolac 30 mg IV every 12 hours
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to assess the efficacy of pentoxifylline in reducing postsurgical complications for breast cancer patients undergoing breast cancer surgery. It aims to evaluate the efficacy of pentoxifylline on postoperative pain and wound healing.

DETAILED DESCRIPTION:
The goal of this clinical trial is to assess the efficacy of pentoxifylline in reducing postsurgical complications for breast cancer patients undergoing mastectomy.

It aims to evaluate the efficacy of adjuvant pentoxifylline in reducing postoperative pain and improving wound healing in breast cancer patients undergoing mastectomy surgery.

Participants will take standard of care treatment with oral pentoxifylline 400 mg 2 hours before surgery, then oral pentoxifylline 400 mg three times per day for 4 weeks, while the control group will only take standard of care. The researchers will compare the difference in pain score and time for wound healing relative to the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients aged 18 to 65 years
2. Patients completed neoadjuvant chemotherapy cycles and scheduled for breast cancer surgery.

Exclusion Criteria:

1. Patients on treatment regimen of phosphodiesterase inhibitors
2. Patients who are taking antiplatelet or anticoagulant treatment
3. Patients who are allergic to phosphodiesterase inhibitors
4. History of recent hemorrhagic events
5. Active peptic ulcer
6. History of psychological problems
7. History of chronic pain management
8. Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative level of pain | 24 hours after surgery
  Postoperative level of pain immediately after the surgery and every 6 hours until 24 hours after surgery using the Numeric Rating Score (NRS) ranging from 0 (indicating no pain) to 10 (expressing the pain as bad as it could possibly be).

SECONDARY OUTCOMES:
Numbers of patients need rescue analgesia | 24 hours after surgery
  The number of patients need rescue analgesia within 24 hours after surgery
Time for wound healing | Within 4 weeks of follow-up after the surgery
  The time for removal of surgical sutures
The incidence of post-surgical complications | Within 4 weeks of follow-up after the surgery
  The incidence of seroma, hematoma, surgical site infection, and skin flap necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Samar A. Dewidar, MSc, Study Chair — clinical pharmacy and pharmacy practice department, Faculty of pharmacy, Mansoura University; Noha O. Mansour, PhD, Study Director — Clinical pharmacy and pharmacy practice department, Faculty of pharmacy, Mansoura University; Moetaza M. Soliman, PhD, Study Director — Clinical pharmacy and pharmacy practice department, Faculty of pharmacy, Mansoura University; Mohamed A. Shams, PhD, Study Director — Clinical pharmacy and pharmacy practice department, Faculty of pharmacy, Mansoura University; Omar H. Abdelaleem, PhD, Principal Investigator — Faculty pf medicine, Mansoura University
Locations (1):
- Oncology center of Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Dewidar SA, Mansour NO, Hamdy O, Elebedy DA, Soliman MM, Shams MEE. Efficacy of using pentoxifylline in patients undergoing breast cancer surgery. Front Pharmacol. 2025 Jul 16;16:1560805. doi: 10.3389/fphar.2025.1560805. eCollection 2025. PMID 40741002